CLINICAL TRIAL: NCT04483115
Title: Multi-center, Randomized，Placebo and Positive Controlled Clinical Study of TPN171H Tablets on Acute Haemodynamics in Patients with Pulmonary Arterial Hypertension
Brief Title: Acute Haemodynamic Study of TPN171H in Patients with Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPN171H-P201
Record Dates: First submitted 2020-07-15; First posted 2020-07-23 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; Acute Haemodynamic Study; PK/PD study; TPN171H; Simmerafil
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- TPN171H 2.5mg group (Experimental): TPN171H 2.5mg tablet + Placebo 10mg tablet
  Interventions: Drug: TPN171H
- TPN171H 5mg group (Experimental): TPN171H 5mg tablet + Placebo 10mg tablet
  Interventions: Drug: TPN171H
- TPN171H 10mg group (Experimental): TPN171H 10mg tablet + Placebo 5mg tablet
  Interventions: Drug: TPN171H
- Placebo group (Placebo Comparator): Placebo 5mg tablet+ Placebo 10mg tablet
  Interventions: Drug: Placebo
- tadalafil 20mg group (Active Comparator): tadalafil tablet 20mg
  Interventions: Drug: Tadalafil
- tadalafil 40mg group (Active Comparator): tadalafil tablets 20mg *2
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: TPN171H — Tablets; Oral; Single dose
  Other Names: Simmerafil
  Arms: TPN171H 10mg group; TPN171H 2.5mg group; TPN171H 5mg group
Drug: Placebo — Tablets; Oral; Single dose
  Arms: Placebo group
Drug: Tadalafil — Tablets; Oral; Single dose
  Other Names: ADCIRCA
  Arms: tadalafil 20mg group; tadalafil 40mg group

SUMMARY:
This study is a phase IIa proof-of-concept study to evaluate the effect of single-dose TPN171H tablets on acute haemodynamic parameters in patients with pulmonary arterial hypertension.The trial is expected to include 60 patients, divided into 6 groups, according to 1:1:1:1:1:1 into the placebo group and the test drugs 2.5mg, 5mg, 10mg group, tadalafil tablets 20mg, 40mg group, each group 10 cases.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, placebo and positive controlled phase IIa proof-of-concept study to evaluate the effect of single-dose TPN171H tablets on acute hemodynamic parameters in patients with pulmonary arterial hypertension.The trial is expected to include 60 patients, divided into 6 groups, according to 1:1:1:1:1:1 into the placebo group and the test drugs 2.5mg, 5mg, 10mg group, tadalafil tablets 20mg, 40mg group, each group 10 cases. During the screening period, the tube placement period, and the observation period, the patients will conduct various inspections and evaluation observations as required.

The Swan-Ganz floating catheter and echocardiography were used to evaluate the efficacy of TPN171H; PK parameters: including Tmax, Cmax, AUC0-t , t1/2,CL/F, Vz/F, λz; Safety evaluation indicators include: vital signs, physical examination, laboratory examination (blood routine, blood biochemistry, blood gas analysis), 12-lead ECG, adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75;
* Patients who have voluntarily decided to participate in this study, and signed the informed consent form;
* Patients who are able to understand and follow study plans and instructions;
* Patients with symtomatic PAH (Group1), a pulmonary vascular resistance (PVR) > 3 Wood, a mean pulmonary artery pressure (mPVP) ≥25 mmHg and a pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg either due to:

  1. Idiopathic PAH (IPAH)
  2. Familial PAH
  3. Associated PAH due to drugs or toxins
  4. Associated PAH due to connective tissue disease
  5. Associated PAH due to congenital heart disease, if patients underwent surgical correction more than 1 year prior to screening
* Have a current diagnosis of being in WHO functional class II or III;
* Patients who are willing to take proper contraceptive during the study and within 3 months after the study completed.

Exclusion Criteria:

* All types of PH except subtypes of Group1 specified in the inclusion criteria;
* Moderate to severe COPD (FEV1 < 60% predicted);
* Moderate to severe restrictive lung disease (FVC < 70% predicted);
* Pre-treatment with PAH therapy within the last 1 months before the screening visit (including endothelin receptor antagonists, PDE5 inhibitors, guanylate cyclase agonist and prostacycline analogues);
* A "positive" response to acute vasodilator testing;
* Coagulation dysfunction (defined as activated partial thromboplastin time and international normalized ratio are both >1.5 times upper limit normal) or patients with potential bleeding risk;
* Hepatic dysfunction indicated by: serum bilirubin>3 times upper limit normal, ALT and AST>2.5 times upper limit normal;
* Renal insufficiency (creatinine clearance<30 mL/min)；
* Systolic blood pressure<90 mmHg at screening;
* QT prolongation at screening, whose values (QTcF) exceeding 450 msec in males and 470 msec in females;
* Have enrolled in/or have a plan of an exercise training program for pulmonary rehabilitation before the screening visit/or during the study;
* Patients who have a recent (within 3 months) history of abusing alcohol or illicit drugs;
* Body weight<40 kg；
* Patients who have participated in a clinical study involving another investigational drug within 1 month before the screening visit;
* For any other reasons that affect compliance with the study protocol, especially the long-term monitoring of floating catheters, according to the decision of investigators;
* HBV, HCV, HIV or Tp infection;
* Patients with gastrointestinal, urinary, reproductive, immunologic, endocrine, or central nervous system disease that, in the opinion of the investigator, will affect the study;
* Have a history of malignancies within 2 years, except for a cured basal cell or skin squamous cell carcinoma;
* Pregnant women, or breast feeding women;
* Patients with hypersensitivity to iloprost or any of the excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of the maximum change in pulmonary vascular resistance(PVR) to the second baseline | Within 24 hours after drug administration

SECONDARY OUTCOMES:
Time of maximum change in PVR | Within 24 hours after drug administration
The area under the curve for reduction in PVR | Within 24 hours after drug administration
Change in arterial oxygenation | Within 24 hours after drug administration
Change in right ventricular function | Within 24 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Principal Investigator — Peking University First Hospital
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital CAMS&PUMC, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - First Affiliated Hospital Of Gannan Medical University, Ganzhou, Jiangxi
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No